CLINICAL TRIAL: NCT01516944
Title: Perioperative Tegafur Gimeracil Oteracil Potassium Capsule Plus Oxaliplatin Versus Capecitabine Plus Oxaliplatin in Patients With Localized Advanced Gastric Cancer
Brief Title: Perioperative Chemotherapy for Potentially Resectable Gastric Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hebei Medical University (Other)
Responsible Party: Principal Investigator, Qun Zhao, Principal Investigator, Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TOTTG030103
Record Dates: First submitted 2012-01-10; First posted 2012-01-25 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Gastric Cancer
Keywords: Tegafur，Gimeracil and Oteracil Potassium Capsules; Capecitabine; Oxaliplatin; perioperative Chemotherapy; Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Tegafur; gimeracil; S 1 (combination); Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- postoperative chemotherapy,SOX (Active Comparator)
  Interventions: Drug: Tegafur, Gimeracil and Oteracil Potassium Capsules；Oxaliplatin
- Perioperative chemotherapy,SOX (Experimental)
  Interventions: Drug: Tegafur, Gimeracil and Oteracil Potassium Capsules；Oxaliplatin
- Perioperative chemotherapy,XELOX (Experimental)
  Interventions: Drug: Oxaliplatin; Capecitabine

INTERVENTIONS:
Drug: Tegafur, Gimeracil and Oteracil Potassium Capsules；Oxaliplatin — Tegafur，Gimeracil and Oteracil Potassium Capsules 80 mg/m2 D1-D14 q3wk and Oxaliplatin 130 mg/m2 D1 q3wk for six cycles postoperation
  Other Names: S-1; Oxaliplatin
  Arms: postoperative chemotherapy,SOX
Drug: Tegafur, Gimeracil and Oteracil Potassium Capsules；Oxaliplatin — Tegafur，Gimeracil and Oteracil Potassium Capsules 80mg/㎡ ,D1-D14 q3wk and Oxaliplatin,130 mg/㎡ D1 q3wk for two cycles preoperation, Tegafur，Gimeracil and Oteracil Potassium Capsules ,80 mg/㎡ D1-D14 q3wk and Oxaliplatin,130 mg/㎡ D1 q3wk for six cycles postoperation
  Other Names: S-1; Oxaliplatin
  Arms: Perioperative chemotherapy,SOX
Drug: Oxaliplatin; Capecitabine — Capecitabine,2000 mg/㎡ D1-D14 q3wk and Oxaliplatin,130 mg/㎡ D1 q3wk for two cycle pre-operation, Capecitabine,2000 mg/㎡ D1-D14 q3wk and Oxaliplatin,130 mg/m2 D1 q3wk for six cycles postoperation
  Other Names: Oxaliplatin; Capecitabine
  Arms: Perioperative chemotherapy,XELOX

SUMMARY:
Stage I：Neoadjuvant therapy

* Tegafur，Gimeracil and Oteracil Potassium Capsules plus oxaliplatin is superior to surgery alone;Capecitabine plus oxaliplatin is non-inferiority to Tegafur，Gimeracil and Oteracil Potassium Capsules plus oxaliplatin

Stage II: Perioperative therapy

* Perioperative Tegafur，Gimeracil and Oteracil Potassium Capsules plus oxaliplatin is superior to adjuvant Tegafur，Gimeracil and Oteracil Potassium Capsules plus oxaliplatin alone;Capecitabine plus oxaliplatin regimen is noninferiority to Tegafur,Gimeracil and Oteracil Potassium Capsules plus oxaliplatin
* A regimen of Tegafur，Gimeracil and Oteracil Potassium Capsules plus oxaliplatin(SOX) and Capecitabine plus oxaliplatin(XELOX) improves survival among patients with incurable locally advanced or metastatic gastric cancer. The investigators assessed whether the addition of a perioperative regimen of SOX or XELOX regimen to adjuvant alone improves R0 resection rate and survival among patients with curable locally advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 -75
* Histologically or cytologically proven in operable advanced gastric adenocarcinoma (including adenocarcinoma of the gastrooesophageal junction)
* ECOG performance status ≦2
* Tumor stage T3/4NxM0
* No distant metastasis (M0)

Exclusion Criteria:

* History of hypersensitivity to fluoropyrimidines, Tegafur，Gimeracil and Oteracil Potassium Capsules , capecitabine, oxaliplatin or the ingredients of this product
* Inadequate hematopoietic function： WBC≦4,000/mm3; ANC≦2,000/mm3; Platelet≦100,000/mm3
* Inadequate organ function which is defined as below:

Total bilirubin >2 pper limit of normal range (ULN); ALT / AST > 2.5 upper limit of normal range (ULN) (>5.0 x ULN if hepatic metastasis); serum creatinine > 1.2 mg/dL, and Ccr > 60 ml/min (estimated by Cockcroft-Gault formulation);

* Symptomatic peripheral neuropathy
* Receiving a concomitant treatment with other fluoropyrimidines
* Pregnancy or lactation women, or women with suspected pregnancy or men unless using a reliable and appropriate contraceptive method.
* Mental status is not fit for chemotherapy therapy presence of serious concomitant illness which might be aggravated by study medication:
* Active cardiac disease e.g. decompensate myocardial infarction within the 6-month period preceding entry into the study.
* History of ventricular arrhythmia or congestive heart failure.
* Significant co-morbid medical conditions, including, but not limited to, Chronic obstructive pulmonary disease, interstitial pneumonia ,pulmonary fibrosis, heart failure, renal failure, hepatic failure, haemorrhagic peptic ulcer, mechanical or paralytic ileus, or poorly controlled diabetes.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 749 (Actual)
Dates: Start 2012-02; Primary Completion 2018-04 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Disease-free survival(DFS) | 3 year

SECONDARY OUTCOMES:
Objective response rate (ORR) | At the end of the study
Disease control rate (DCR) | At the end of the study
  To Assess disease control rate (DCR) as defined CR + PR + SD assessed by RECIST criteria
Down staging rate | Within 3 weeks after surgery
  After the pathological examination of resected specimen
Overall survival (OS) | 5 year
Adverse events | Side effects during observation
  Investigators graded all adverse events and toxic effects according to the National Cancer Institute's Common Toxicity Criteria, version 2.0. The number of Participants with adverse events will be recorded at each treatment visit.
R0-resection rate | Within 3 weeks after surgery
  After the pathological examination of resected specimen

CONTACTS AND LOCATIONS:
Overall Officials: Qun Zhao, Doctor, Principal Investigator — Hebei Medical University
Locations (1):
- Department of General Surgery, Shijiazhuang, Hebei, China

REFERENCES:
- [Derived] Ding P, Wu J, Wu H, Sun C, Meng M, Lowe S, Tian Y, Guo H, Meng L, Zhao Q. Comment on 'Hand grip strength-based cachexia index as a predictor of cancer cachexia and prognosis in patients with cancer' by Xie et al. J Cachexia Sarcopenia Muscle. 2023 Oct;14(5):2449-2451. doi: 10.1002/jcsm.13298. Epub 2023 Jul 28. No abstract available. PMID 37501640
- [Derived] Zhao Q, Lian C, Huo Z, Li M, Liu Y, Fan L, Tan B, Zhao X, Zhang Z, Wang D, Liu Y, Guo H, Yang P, Tian Y, Li Y. The efficacy and safety of neoadjuvant chemotherapy on patients with advanced gastric cancer: A multicenter randomized clinical trial. Cancer Med. 2020 Aug;9(16):5731-5745. doi: 10.1002/cam4.3224. Epub 2020 Jun 24. PMID 32583567